CLINICAL TRIAL: NCT06098196
Title: Effects of Aminophylline Bolus on Eleveld and Schnider TCI (Target Controlled Infusion) Concentrations at Return of Responsiveness and on BIS (Bispectral Index) After Total Intravenous Anaesthesia With TCI
Brief Title: Effects of Aminophylline Bolus on TCI (Target Controlled Infusion) Concentrations at Return of Responsiveness
Acronym: TCI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal investigator, University of Padova
Other Study IDs: Teoawake
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Propofol; Anesthesia Brain Monitoring
MeSH Terms: interventions — Aminophylline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aminophylline: Patients who received Aminophylline bolus (4 mg/kg) at the end of general anesthesia conducted with Eleveld or Schnider TCI model (this model was chosen at anesthesiologist's discretion)
  Interventions: Drug: Aminophyllin
- Not Aminophylline: Patients who did not received Aminophylline bolus (4 mg/kg) at the end of general anesthesia conducted with Eleveld or SchniderTCI model (this model was chosen at anesthesiologist's discretion
  Interventions: Drug: Aminophyllin

INTERVENTIONS:
Drug: Aminophyllin — Patients will be observationally included in the Elveld TCI or Schnider TCI group and recevied or not Aminiophylline bolus. The TCI model, such as the aminophylline delivery or not, is chosen at anesthesiologist's discretion, as suggested in literature

SUMMARY:
Aminophylline is an intravenous drug commonly utilized for asthma. However, some preclinical studies and few case reports and case series have described its utility in decrease the timing of return of consciousness after Propofol anaesthesia with an intravenous bolus of 4 mg/kg.

We aimed to compare its effect during a total Intravenous Anaesthesia with Target Controlled Infusion (TIVA-TCI) routinely utilized for general anaesthesia in our hospital.

DETAILED DESCRIPTION:
Aminophylline is an intravenous drug commonly utilized for asthma. However, some preclinical studies and few case reports and case series have described its utility in decrease the timing of return of consciousness after Propofol anaesthesia with an intravenous bolus of 4 mg/kg.

We aimed to compare its effect during a total Intravenous Anasethesia with Target Controlled Infusion (TIVA-TCI) routinely utilized for general anaesthesia in our hospital (with Eleveld or Schnider Pharmacokinetic/Pharmacodynamic-PK/PD model).

The timing from stop of propofol infusion to eye opening and return of responsiveness, the relative Concentration of Propofol (CeP) and the power spectrum of the Bispectral Index (BIS) with or without aminophylline bolus were taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol (Eleveld or Schnider model) and Remifentanil (Minto model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and Remifentanil TCI, with or without aminophylline bolus at the end of surgery will be recruited
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Correlation between Concentration at the effector site of Propofol after Aminophylline | We will collected data about Drugs concentration and BIS values during general anaesthesia. We will collect BIS and TCI Propofol values during all the duration of anesthesia, form the start of anaesthesia until the emergence from anesthesia
  Discover if, after an aminophylline bolus, there are differences between Concentrations at the effector site and timing at eye opening of Propofol using the Eleveld TCI model or Schnider TCI model, after standard general anaesthesia conducted with Propofol and remifentanil delivered with target controlled infusion pumps, usually adopted in our Hospital to delivery general anaesthesia

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - ULSS 2 Marca Trevigiana, Treviso, Tv
  - ULSS2 Marca Trevigiana, Treviso

IPD SHARING:
Plan to Share IPD: Undecided